CLINICAL TRIAL: NCT06838195
Title: A Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial Evaluating the Protective Efficacy, Immunogenicity, and Safety of the S. Flexneri-S. Sonnei Bivalent Conjugate Vaccine in Infants and Children Aged 6 Months to 5 Years in Bangladesh
Brief Title: Clinical Trial of the S. Flexneri-S. Sonnei Bivalent Conjugate Vaccine
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PR-24079
Record Dates: First submitted 2025-02-07; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Dysentery; Dysentery, Shigella
Keywords: S. Flexneri-S. Sonnei bivalent conjugate vaccine
MeSH Terms: conditions — Dysentery; Dysentery, Bacillary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaccine group (Experimental): 4000 subjects aged 6 months to 5 years are enrolled in this group.
  Interventions: Biological: S. Flexneri-S. Sonnei bivalent conjugate vaccine
- Placebo group (Placebo Comparator): 4000 subjects aged 6 months to 5 years are enrolled in this group.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: S. Flexneri-S. Sonnei bivalent conjugate vaccine — Subjects receive two doses of the vaccine on the day of randomisation (day 0) and day 30.
  Arms: Vaccine group
Biological: Placebo — Subjects receive two doses of the placebo on the day of randomisation (day 0) and day 30.
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to evaluate the protective efficacy of S. Flexneri-S. Sonnei bivalent conjugate vaccine against diarrhea caused by Shigella infection in infants and children aged 6 months to 5 years. Researchers will observe the incidence of diarrhea of any severity due to Shigella flexneri and Shigella sonnei infection 30 days after full immunization. The subjects will receive 2 doses of vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children aged 6 months to 5 years.
* Legal guardians voluntarily agree to participate in the study and sign an informed consent form.
* Legal guardians agree to comply with the requirements of the clinical trial protocol and are willing and able to participate in all planned follow-ups.
* The subject's guardian agrees that the subject should not abuse antibiotics. If needed，antibiotics should be used under the guidance of a doctor and avoid taking antibiotics on their own during the clinical trial.
* Based on medical history, physical examination, and the investigator's judgment, the subject is determined to be in good health.

Exclusion Criteria:

* History of confirmed bacterial dysentery in the past 6 months.
* Serious allergy to tetanus toxoid, history of severe allergies, fever above 39.5°C following previous vaccination with a prophylactic biological product.
* Currently suffering from serious intestinal diseases, symptoms of diarrhea, abdominal pain, or bloody purulent stools in the past 15 days.
* Diagnosed pathological jaundice currently.
* Confirmed diagnosis of thrombocytopenia or other coagulation disorders.
* Known or suspected immunological deficiencies (e.g., perianal abscesses indicating potential immune deficiency in infants and young children), long-term treatment (≥14 days) with immunosuppressants within half a year before vaccination (radiotherapy, chemotherapy, systemic corticosteroids ≥2 mg/kg/day, antimetabolites, cytotoxic drugs), or parents confirmed to have HIV infection.
* Receipt of immunoglobulins/blood products (except hepatitis B immunoglobulin) within 3 months before vaccination.
* Severe congenital anomalies (important organ function impairment), severe malnutrition, developmental disorders, severe hereditary diseases.
* Currently suffering from the following diseases:

  1. Severe liver or kidney diseases, cardiovascular diseases, malignant tumors, and other severe chronic diseases.
  2. Diagnosed serious infectious diseases, such as tuberculosis, viral hepatitis, etc.
  3. Severe asthma.
  4. Generalized rashes, dermatophytosis, skin suppuration, or blistering.
  5. Convulsions, epilepsy, encephalopathy, psychiatric disorders or family history of psychiatric disorders.
* Planning to participate or currently participating in other vaccine or drug clinical trials.
* Any condition that the investigators believe may affect the evaluation of the study.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8000 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2028-07-02 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
The protective efficacy of S. Flexneri-S. Sonnei bivalent conjugate vaccine | From day 30 post full immunization to the subsequent 24-month period.
  The efficacy will be assessed by comparing the incidence rate of laboratory-confirmed S. flexneri-associated or S. sonnei-associated diarrhea between the vaccinated group and the placebo group.
  Statistical Analysis:
  Protective efficacy(%)=(control group incidence (person-year incidence)- vaccine group incidence (person -year incidence))/control group incidence (person-year incidence)x100%

SECONDARY OUTCOMES:
The protective efficacy against diarrhea cases with positive bacterial culture for Shigella species | From he first dose of immunization to 24-month period post full immunization.
  Evaluation of the protective efficacy of the vaccine against diarrhea cases with positive bacterial culture for Shigella species.
Positive PCR testing for Shigella species | From day 30 post full immunization to the subsequent 24-month period.
  Evaluation of diarrhea cases with positive PCR testing for Shigella species
IgG antibody seroconversion (fourfold increase) rate on day 30 post full immunization for subgroup 1. | The 30th day after two doses of the vaccine.
  Subjects in immunogenicity subgroup 1, vaccine serotype-specific Shigella flexneri and Shigella sonnei IgG antibody seroconversion (fourfold increase) rate on day 30 post full immunization.
IgG antibody concentration on day 30 post full immunization for subgroup 1. | The 30th day after two doses of the vaccine.
  For subjects in immunogenicity subgroup 1, vaccine serotype-specific Shigella flexneri and Shigella sonnei antibody concentration on day 30 post full immunization.
IgG antibody seroconversion (fourfold increase) rate on day 30 post full immunization for subgroup 2. | From 30 day to 1 year after the first immunization.
  For subjects in immunogenicity subgroup 2, vaccine serotype-specific Shigella flexneri and Shigella sonnei IgG antibody seroconversion (fourfold increase) rate on day 30 post the first dose, day 30 post full immunization, half a year after the first immunization, and one year after the first immunization.
IgG antibody concentration on day 30 post full immunization for subgroup 2. | From 30 day to 1 year after the first immunization.
  For subjects in immunogenicity subgroup 2, vaccine serotype-specific Shigella flexneri and Shigella sonnei antibody concentration on day 30 post the first dose, day 30 post full immunization, half a year after the first immunization, and one year after the first immunization.
AEs within 0-30 minutes after vaccination | Within 30 minutes after each dose of vaccine
  The occurrence of any adverse events within 30 minutes after each dose of vaccine (number of instances, number of cases, incidence rate, and the relationship to the vaccine administration)
Solicited AEs within 0-7 days after vaccination | Within 0-7 days after each vaccine dose.
  The occurrence of solicited adverse events from Day 0 to Day 7 after each vaccine dose (number of instances, number of cases, incidence rate, and the relationship to the vaccine administration)
Unsolicited AEs within 0-30 days after vaccination | Within 0-30 days after each vaccination
  The occurrence of unsolicited adverse events from Day 0 to Day 30 after each vaccine dose (number of instances, number of cases, incidence rate, and the relationship to the vaccine administration).
SAE within 0-6 months after primary immunization | Within 0-6 months after primary immunization.
  The occurrence of Serious Adverse Events (SAEs) from after the first dose to 6 months after complete immunization (number of instances, number of cases, incidence rate, and the relationship to the vaccine administration)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Du, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Icddr,B, Dhaka, Bangladesh